CLINICAL TRIAL: NCT04614727
Title: Desensitizing Efficacy of Polymeric Nano Calcium Fluoride Containing Varnish Versus Casein Phosphopeptide Amorphous Calcium Phosphate Containing Fluoride Varnish: Randomized Clinical Trial
Brief Title: Desensitizing Efficacy of Polymeric Nano Calcium Fluoride Containing Varnish
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samar Saad (Other)
Responsible Party: Sponsor-Investigator, Samar Saad, principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Polymeric Nano Calcium Fluorid
Record Dates: First submitted 2020-10-23; First posted 2020-11-04 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin sensitivity ,nano calcium fluoride, nano fluorapatite,Casein Phosphopeptide Amorphous Calcium Phosphate.
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- polymeric nano calcium fluoride containing varnish, NANO SEAL. (Experimental)
  Interventions: Combination Product: polymeric nano calcium fluoride containing varnish NANO SEAL
- Casein Phosphopeptide Amorphous Calcium Phosphate Containing Fluoride Varnish,MI varnish (Other): CPP-ACP with 5%NaF
  Interventions: Combination Product: polymeric nano calcium fluoride containing varnish NANO SEAL

INTERVENTIONS:
Combination Product: polymeric nano calcium fluoride containing varnish NANO SEAL — It consists of four components Silicone polymer provides excellent adhesion to enamel and dentine, with transparent formula. NANO-fluoroapatite flows into enamel micro cracks & seals it, penetrating into the dentinal tubules closing them eventually. As for the NANO-calcium fluoride it behaves as a fluoride reservoir, provides gradual and long-term fluoride release. The fourth component Amine fluoride (Olaflur) provides immediate fluoride ion release and accelerates natural remineralization.

SUMMARY:
The aim of this study is to evaluate the Desensitizing efficacy of polymeric nano calcium fluoride containing varnish and its implementation into clinical practice.

DETAILED DESCRIPTION:
Increasing the demand to find a desensitizing agent that should be biocompatible, easy to apply, painless, not changing the dental color, fast onset, and maintain a long-term effect gives a highlight to the patented formula of the polymeric nano calcium fluoride which newly introduced into the practice .

OliNano SEAL is an innovative "varnish-like" protector based on a patented silicone polymer with a true nano technology that provides an exceptional adhesion to enamel and dentin without prior etching for approximately 12 months (other available products max. 2-3 months).

It consists of four components Silicone polymer provides excellent adhesion to enamel and dentine, with transparent formula. NANO-fluoroapatite flows into enamel micro cracks & seals it, penetrating into the dentinal tubules closing them eventually. As for the NANO-calcium fluoride it behaves as a fluoride reservoir, provides gradual and long-term fluoride release. The fourth component Amine fluoride (Olaflur) provides immediate fluoride ion release and accelerates natural remineralization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene.
* The age range of 18-65 years.
* Patients from both gender.
* Patients suffering from pain due to dentin hypersensitivity.
* hypersensitive areas on facial surfaces of the teeth (incisors, cuspids, bicuspids, and first molars with exposed cervical dentine).
* non carious cervical lesions: abrasion,erosion, abfraction, and recession with cervical dentin exposure

Exclusion Criteria:

* Patient with bad oral hygiene.
* Patients with constant use of analgesic, antihistaminic, anticonvulsive, sedative, tranquilizing, or anti-inflammatory medications 72 hours before treatment and pain assessment.
* patients having received any desensitizing treatment during the last 3 months.
* Patients with allergy of any materials will be used in the study . teeth with pulpitis.
* teeth with periodontal disease installed.
* teeth exhibiting mobility (grade 2 or 3).
* carious lesions, fractured teeth, defective restorations or prosthesis.
* Patients with orthodontics appliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-10 (Estimated); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale VAS | six months
  from 0-10 Pain absent: 0 Low pain:(1-3) Moderate pain: (4-6) Intense pain: (7-9) Extremely intense pain: 10.
Schiff air score | six months
  from 0-3 0: Tooth/subject did not respond to the air stimulus.
  1. Tooth/subject responded to the air stimulus but did not request discontinuation of the stimulus.
  2. Tooth/subject responded to the air stimulus and requested discontinuation or moved from the stimulus.
  3. Tooth/subject responded to the air stimulus, considered the stimulus to be painful, and requested discontinuation.

SECONDARY OUTCOMES:
Dentinal tubule occlusion | six months
  Fully open, partially occluded and fully occluded dentinal tubules. (Percentage %)

IPD SHARING:
Plan to Share IPD: Yes